CLINICAL TRIAL: NCT05185921
Title: Effectiveness of Virtual Cognitive Behavioral Therapy(CBT) on the Quality of Life of HIV-infected Persons, COVID-19, With Anxiety and Depression, 2021-2022.
Brief Title: CBT and Quality of Life of People With HIV, COVID-19 and Anxiety or Depression
Acronym: COVIHMENT-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Peruana Cayetano Heredia (Other)
Collaborators: Hospital Nacional Alberto Sabogal Sologuren (Other); University of Minnesota (Other)
Responsible Party: Principal Investigator, Pavel Jaime Contreras Carmona, Principal Investigator, Universidad Peruana Cayetano Heredia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 207454
Record Dates: First submitted 2022-01-06; First posted 2022-01-11 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Quality of Life; Anxiety; Depression
Keywords: HIV; COVID-19; Cognitive Behavioral Therapy
MeSH Terms: conditions — Anxiety Disorders; Depression; COVID-19

STUDY DESIGN:
Intervention Model Description: 182 patients selected by simple randomization from a list of people at the Health Center who meet the eligibility criteria will be divided at study enrollment into an intervention group (n=91) and a control group (n=91). Assignment to each group will be 1:1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive-behavioral therapy virtual (Experimental): The intervention will be provided by 2 psychotherapists. The total of sessions will be eight carried out weekly, for 2 to 3 months. They will also receive standard treatment, i.e. psychiatric management with or without drugs.
  Interventions: Behavioral: Trial-based Cognitive therapy
- Control (No Intervention): They will only receive standard treatment, i.e. psychiatric management with or without drugs.

INTERVENTIONS:
Behavioral: Trial-based Cognitive therapy — The virtual CBT will be provided by 02 psychotherapists, who will follow a protocol developed for this study. The number of sessions will be eight, which will be held weekly, projecting an intervention time of 2 to 3 months considering the possibility of rescheduling any of the sessions for reasons derived from the participant People with relevant cognitive impairment that prevents them from answering the questionnaire questions or providing informed consent are excluded.
  Arms: Cognitive-behavioral therapy virtual

SUMMARY:
Experimental open-label randomized clinical trial to determine the effect of virtual Cognitive Behavioral Therapy (CBT) on the quality of life of patients with HIV, COVID-19 and anxiety or depression. It will be carried out at the hospital for 6 months, where people over 18 years of age with HIV from the infectious disease service will participate.

In the study, patients will be randomized 1:1 in an intervention group, who will receive eight sessions of virtual CBT by 02 psychotherapists, and a control group. Additionally, patients will be consulted about the participation of at least one adult family member or caregiver in the study, if the patient and the family member agree, the family member or caregiver will enter the study.

The informed consent process will be conducted by telephone, during the call the recruiting staff will read the consent document and the participant (patient and family member or caregiver) will give their consent by answering affirmatively to the questions asked at the end of the document. The main objective will be evaluated by comparing the quality of life measurement at three months with the baseline measurement, as well as the variation of anxiety and depression scores.

DETAILED DESCRIPTION:
Introduction: Confrontational measures such as social isolation and confinement due to the COVID-19 pandemic and the experience of illness have affected people's emotional health by generating or exacerbating anxious and depressive symptoms. This effect may be magnified in people with HIV, contributing to the deterioration of their quality of life.

Objective: To determine the effect of virtual Cognitive Behavioral Therapy on the quality of life of patients with HIV, COVID-19, and anxiety or depression of Social Security.

Design: Experimental open-label randomized clinical trial. To be conducted at the hospital during 6 months.

Materials and Methods:

Participants will be over 18 years of age with HIV from the infectious disease service of the hospital selected for this study. Quality of life, depression, anxiety, multimorbidity and post COVID-19 symptoms will be evaluated. Data will be collected by telephone calls and online questionnaires. Data will be recorded using Redcap online software. To evaluate the effect of virtual cognitive behavioral therapy measured at 4 months, McNemar's Chi-square tests will be used for categorical dependent variables and Student's t-tests for related samples in the case of numerical dependent variables using STATA v. 17.0 statistical software.

Ethical aspects:

The study will be reviewed by the hospital services and the institutional ethics committee. The confidentiality of each participant's information will be maintained through codes that do not allow patient identification.

ELIGIBILITY:
Inclusion Criteria:

* Patients affiliated with Social Security.
* HIV patients diagnosed with COVID-19, anxiety or depression.
* Have a telephone to contact them.
* Family member or adult caregiver of the patient selected for the study and who previously authorized the invitation to the family member or caregiver to participate in the study.

Exclusion Criteria:

* Difficulty to read and to write
* Being currently in psychotherapy
* Clinical diagnoses of neurocognitive or psychotic disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Change in Quality of life | Baseline, after 1 and 3 month
  Quality of life will be assessed with the Spanish 5-dimensional quality of life questionnaire (EQ-5D-3L). This questionnaire can be used in the general population and essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'. The VAS can be used as a quantitative measure of health outcome that reflects the patient's own judgement.

SECONDARY OUTCOMES:
Change in Anxiety | Baseline, after 1 and 3 month
  This condition will be evaluated with the seven-question Generalized Anxiety Disorder (GAD-7), in its Spanish version and with a dichotomous categorization, as well as according to the level of severity. This questionnaire uses a 4-point Likert scale from 0 to 3, with a total score ranging from 0 to 21 points, the higher the score, the greater the degree of anxiety. A score higher than 10 is considered as anxiety.
Change in Depression | Baseline, after 1 and 3 month
  This condition will be evaluated using the Patient Health Questionnaire (PHQ-9), a depression scale in its Spanish version, with a dichotomous categorization, as well as according to the level of severity. This nine-question scale awards one point for each response indicating depressive symptoms; the higher the score, the greater the presence of depressive symptoms; from 0 to 4 points is considered normal, mild from 5 to 8 points, moderate from 9 to 10 points and severe from 12 to 15 points.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Nacional Alberto Sabogal Sologuren, Lima, Peru

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Major depressive disorder and its association with adherence to antiretroviral therapy and quality of life: cross-sectional survey of people living with HIV/AIDS in Northwest Ethiopia — https://bmcpsychiatry.biomedcentral.com/articles/10.1186/s12888-020-02865-w
- See also: Magnitude and predictors of common mental disorder among people with HIV/AIDS in Ethiopia: a systematic review and meta-analysis — https://bmcpublichealth.biomedcentral.com/articles/10.1186/s12889-020-08800-8
- See also: Internet-Delivered Cognitive Behavioural Therapy for Major Depression and Anxiety Disorders: A Health Technology Assessment — https://pubmed.ncbi.nlm.nih.gov/30873251/
- See also: The Role of Telehealth in Reducing the Mental Health Burden from COVID-19 — https://pubmed.ncbi.nlm.nih.gov/32202977/